CLINICAL TRIAL: NCT06613217
Title: A Phase 1 Study of Oral PCLX-001 in Relapsed/Refractory (R/R) Acute Myeloid Leukemia (AML)
Brief Title: Study of Oral PCLX-001 in R/R Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pacylex Pharmaceuticals (Industry)
Collaborators: Ozmosis Research Inc. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PCLX-001-02
Record Dates: First submitted 2024-08-01; First posted 2024-09-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Relapsed Adult AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- zelenirstat intervention in R/R AML at 40mg daily (Experimental): Three patients will be treated at 40 mg daily dose level. If 0/3 patients experience DLT, 3 patients will be treated at the next dose level.
  Interventions: Drug: zelenirstat
- zelenirstat intervention in R/R AML at 70mg daily (Experimental): Three patients will be treated at 70 mg daily dose level. If 0/3 patients experience DLT, 3 patients will be treated at the next dose level.
  Interventions: Drug: zelenirstat
- zelenirstat intervention in R/R AML at 100mg daily (Experimental): Three patients will be treated at 100 mg daily dose level. If 0/3 patients experience DLT, 3 patients will be treated at the next dose level.
  Interventions: Drug: zelenirstat
- zelenirstat intervention in R/R AML at 140mg daily (Experimental): Three patients will be treated at 140 mg each dose level. If 0/3 patients experience DLT, 3 patients will be treated at the next dose level.
  Interventions: Drug: zelenirstat
- zelenirstat intervention in R/R AML at 210mg daily (if needed) (Experimental): Three patients will be treated at 210 mg daily dose level. If 0/3 patients experience DLT, 3 patients will be treated at the next dose level.
  Interventions: Drug: zelenirstat
- zelenirstat intervention in R/R AML at 280mg daily (if needed) (Experimental): Three patients will be treated at 280 mg daily dose level. If 0/3 patients experience DLT, 3 additional patients will be treated at the same dose and the study will be concluded.
  Interventions: Drug: zelenirstat

INTERVENTIONS:
Drug: zelenirstat — Zelenirstat will be administered orally, once daily, on 28-day cycles, at the same time each day.
  Other Names: PCLX-001

SUMMARY:
This is a dose-finding study of oral zelenirstat (PCLX-001) in patients with R/R AML. There are two parts to the study: Dose Escalation and Dose Expansion.

DETAILED DESCRIPTION:
This is a dose-finding study of oral PCLX-001 in patients with R/R AML. There are two parts to the study: Dose Escalation and Dose Expansion.

Dose Escalation will determine the minimum safe and biologically-effective dose of daily oral PCLX-001 in patients with R/R AML. The Bayesian optimal interval (BOIN) design will be used for dose escalation, informed by real-time assessment of safety, efficacy, PK and PD in each dose cohort. A maximum of 15 patients will enroll in the dose escalation part. Oral PCLX-001 will be provided as continuous daily dosing on a 28-day cycle. The starting dose will be 40 mg. AML patients will be evaluated for toxicity, PK, and the relationship between PK observed in this AML trial with universally co-administered CYP3A inhibitor drugs (as in this setting, azole antifungals are continuously administered to this population), in comparison with PK data derived from patients with NHL and solid tumors without co-administered CYP3A inhibitors. These data will be integrated to inform the decision on the minimum safe and biologically-effective dose to be used in the expansion cohort.

PCLX-001 will be administered as an oral daily dose on a 28-day cycle as per the dose level schedule below.

Dose Escalation Schedule: (1 cycle = 28 days)

1. Daily oral dose of 40mg
2. Daily oral dose of 70mg
3. Daily oral dose of 100mg
4. Daily oral dose of 140mg
5. Daily oral dose of 210mg
6. Daily oral dose of 280mg

Trial will start at 40mg based on results from an ongoing independent dose escalation trial in NHL and solid tumors. If DLT is not observed at the dose of 280 mg, this dose will be considered the minimum safe and biologically-effective dose to be used in the expansion cohort.

Dose expansion. 20 evaluable patients will be accrued and treated with the minimum safe and biologically-effective dose. PCLX-001 will be administered as an oral daily dose on a 28-day cycle to determine the safety and preliminary clinical activity of PCLX-001.

Dosing Administration PCLX-001 will be administered orally, once daily, on 28-day cycles, at the same time each day.

ELIGIBILITY:
Inclusion Criteria:

-

The following inclusion criteria apply to ALL (dose escalation and dose expansion) patients:

1. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained before any study-specific procedures are performed.
2. Male or female patients aged ≥ 18 years
3. A diagnosis of AML as per 2016 WHO classification (Arber et al, 2016)
4. Patients must have received at least one prior therapy for AML
5. Patient must not be eligible for other therapies expected to provide clinical benefit
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (Appendix A).
7. The use of chemotherapeutic or anti-leukemic agents is not permitted during the study with the following exceptions: (1) intrathecal (IT) therapy for patients with controlled CNS leukemia at the discretion of the Investigator. Controlled CNS leukemia is defined by the absence of active clinical signs of CNS disease and no evidence of CNS leukemia on the most recent 2 simultaneous cerebrospinal fluid (CSF) evaluations. (2) Use of hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy. These medications will be recorded in the case-report form.
8. Patients must have adequate liver function as assessed by the following laboratory tests to be conducted within 7 (±3) days before the first dose of study drug:

   1. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) unless increase is due to hemolysis or congenital disorder such as Gilbert's syndrome
   2. ALT and AST ≤ 2.5 times ULN or ≤ 5 times ULN for patients with malignant liver involvement
9. Patients must have adequate kidney function, as assessed by both:

   1. the estimated glomerular filtration rate (eGFR) >60 mL/min within 7 (±3) days before the first dose of study drug (eGFR to be calculated by the Cockcroft-Gault formula)
   2. creatinine ≤ 1.5 times the ULN
10. Adequate cardiac function per institutional normal measured by echocardiography or multi-gated acquisition (MUGA) scan (Left ventricular ejection fraction (LVEF) ≥ 50%)
11. Ability to take oral medication
12. Women of childbearing potential must have a negative serum beta human chorionic gonadotropin (β- human chorionic gonadotropin (HCG)) pregnancy test obtained within 7 (±3) days before the start of administration of study drug.

    a. Note: A woman is of childbearing potential, i.e., fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy.
13. Women of childbearing potential and fertile men must agree to use adequate contraception when sexually active from signing of the informed consent form for the full study until at least 6 months after the last study drug administration. Patients must agree to utilize 2 reliable and acceptable methods of contraception simultaneously. A man is considered fertile after puberty unless permanently sterile by bilateral orchiectomy. Men being treated with PCLX-001 are advised not to father a child during and up to 6 months after treatment; prior to treatment, advice should be sought for conserving sperm due to the chance of irreversible infertility as a consequence of treatment with PCLX-001. Female partners of childbearing potential from male study participants have to use adequate contraception / birth control between signing of the informed consent and 6 months after the last administration of the study drug if the male study participant is not sterilized. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control. Highly effective (failure rate of less than 1% per year) contraception methods, when used consistently and correctly, include:

    1. Combined (estrogen and progestin containing: oral, intravaginal transdermal and progestin-only (oral, injectable, implantable) hormonal contraception associated with inhibition of ovulation.
    2. Intra-uterine device (IUD) or intrauterine hormone-releasing system (IUS).
    3. Bilateral tubal occlusion or vasectomized partner (provided that partner is the sole sexual partner and has received medical assessment of the surgical success).
    4. Sexual abstinence (reliability to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient).
14. Male patients with a female partner of reproductive potential must use a condom and ensure that an additional form of contraception is also used during treatment and until 6 months after last study drug administration. Patients must agree to utilize reliable and acceptable methods of contraception simultaneously.

Exclusion Criteria:

-

The following exclusion criteria apply to ALL (dose escalation and dose expansion) patients:

1. Acute promyelocytic leukemia.
2. Known hypersensitivity to the study drugs or excipients of the preparations or any agent given in association with this study
3. History of cardiac disease: congestive heart failure New York Heart Association (NYHA) class > II, unstable angina (angina symptoms at rest), new-onset angina (within the past 6 months before study entry), myocardial infarction within the past 6 months before study entry, or uncontrolled cardiac arrhythmias
4. Uncontrolled arterial hypertension despite optimal medical management (per investigator's opinion)
5. Moderate or severe hepatic impairment, i.e., Child-Pugh class B or C
6. Known HIV infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA load, CD4+ counts/levels > 250, no history of AIDs-defining opportunistic infection within the past 12 months, and stable for at least 4 weeks on same anti-HIV retroviral medications.
7. Patients who have an active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection requiring treatment. Patients with chronic HBV or HCV infection are eligible at the investigator's discretion provided that the disease is stable and sufficiently controlled under treatment.
8. Infections of CTCAE Grade 2 not responding to therapy or active clinically serious infections of CTCAE Grade > 2
9. Uncontrolled seizure disorder requiring therapy with strong CYP3A4 inducers such as carbamazepine and phenytoin
10. Previous or concurrent cancer that is distinct in primary site or histology from AML, with the exception of the following previous or concurrent cancer types:

    1. Curative treatment for localized cancer completed without signs of recurrence and treatment-related toxicity and low risk of recurrence as assessed by the investigator,
    2. In-situ prostate cancer, Gleason Score <7, prostate-specific antigen <10 ng/mL (very low risk and low risk, according to therapy guidelines, e.g., the National Comprehensive Cancer Network guideline; active surveillance / observation is a recommended option).
11. Inability to swallow oral medications
12. Any malabsorption condition that may significantly alter the absorption of PCLX-001.
13. Breastfeeding. Female patients must not breastfeed during treatment and until 4 months after last study drug administration.
14. Acute toxic effects (CTCAE Grade ≥2) of previous anticancer chemotherapy or immunotherapy that have not yet stabilized or if significant post-treatment toxicities have been observed. (Note however that toxic effects of previous anticancer therapy considered as chronic, such as chemotherapy-induced neuropathy, fatigue, alopecia, or anorexia of CTCAE Grade <2, for which further resolution is not expected, do not prevent participation in this study.)
15. Patients on active radiation therapy or active antineoplastic therapy for a concurrent malignancy at the time of screen. Maintenance therapy, hormonal therapy, or steroid therapy for well-controlled malignancy is allowed.
16. Previous assignment to treatment during this study
17. Concomitant participation in another clinical study with investigational medicinal product(s)
18. Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
19. Clinically relevant findings in the ECG such as a second- or third-degree atrioventricular block, prolongation of the QRS complex > 120 ms (except for bundle branch block pattern), or prolongation of the of the QTc interval (Fridericia) over 450 ms unless agreed otherwise between the investigator and the sponsor's medically responsible person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
To determine, during the dose escalation phase, the recommended dose of zelenirstat for the dose expansion phase of the trial. | Up to 18 months
  The recommended dose will be the dose level below that for the cohort in which maximum tolerated dose (MTD) was reached/exceeded. MTD will have been reached when 2 or more patients in a cohort experience DLT.

SECONDARY OUTCOMES:
To evaluate the clinical response rate in patients treated with zelenirstat with AML. | Up to 18 months
  Tumor response and progression of AML will be evaluated by the investigator at each study center.

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Pemmaraju, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Centre, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beauchamp E, Yap MC, Iyer A, Perinpanayagam MA, Gamma JM, Vincent KM, Lakshmanan M, Raju A, Tergaonkar V, Tan SY, Lim ST, Dong WF, Postovit LM, Read KD, Gray DW, Wyatt PG, Mackey JR, Berthiaume LG. Targeting N-myristoylation for therapy of B-cell lymphomas. Nat Commun. 2020 Oct 22;11(1):5348. doi: 10.1038/s41467-020-18998-1. PMID 33093447
- [Background] Sangha R, Davies NM, Namdar A, Chu M, Spratlin J, Beauchamp E, Berthiaume LG, Mackey JR. Novel, First-in-Human, Oral PCLX-001 Treatment in a Patient with Relapsed Diffuse Large B-Cell Lymphoma. Curr Oncol. 2022 Mar 13;29(3):1939-1946. doi: 10.3390/curroncol29030158. PMID 35323358
- [Result] Beauchamp E, Gamma JM, Cromwell CR, Moussa EW, Pain R, Kostiuk MA, Acevedo-Morantes C, Iyer A, Yap M, Vincent KM, Postovit LM, Julien O, Hubbard BP, Mackey JR, Berthiaume LG. Multiomics analysis identifies oxidative phosphorylation as a cancer vulnerability arising from myristoylation inhibition. J Transl Med. 2024 May 7;22(1):431. doi: 10.1186/s12967-024-05150-6. PMID 38715059